CLINICAL TRIAL: NCT01655719
Title: Phase 2 Study of Pioglitazone in Thyroid Cancers That Contain the PAX8-PPARgamma Fusion Gene
Brief Title: Pioglitazone in Thyroid Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald J. Koenig, MD PhD, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011.097; R01CA166033 (NIH)
Record Dates: First submitted 2012-07-25; First posted 2012-08-02 (Estimated); Results first posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Thyroid Cancers That Contain the PAX8-PPARgamma Fusion Gene
MeSH Terms: interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pioglitazone Treatment (Experimental): If eligible, subjects can participate in 1 or both parts of this study as follows:
  Part 1: In the initial main portion of the study subjects will receive 24 -28 weeks of therapy with pioglitazone at the dosage approved for the control of diabetes. Response will be evaluated per RECIST. Safety measure are outlined in the protocol including weekly weigh ins, calls, labs, exams, etc.
  Part 2: A secondary protocol is then available to subjects who complete the main initial study with less than complete response per RECIST. They can undergo a radioiodine scan to see if the treatment with pioglitazone has sensitized their disease to radioiodine. If it has - they can pursue the radioiodine treatment.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone
  Other Names: Actos

SUMMARY:
Through this trial the investigators hope to learn if a drug, Actos (pioglitazone), is useful in treating a certain kind of metastatic thyroid cancer. Actos is approved by the FDA to treat diabetes. It has not been approved by the FDA to treat cancer, so its use in this study is considered experimental.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed thyroid carcinoma with the PAX8-PPARgamma translocation (translocation testing will be performed on archived tissue during the screening period).

   Refractory to radioactive iodine (RAI) as defined by: the tumor does not concentrate RAI; or the patient has had RAI within the last 16 months and has had progression despite that RAI; or the last RAI treatment was >16 months ago and the patient progressed after at least two RAI treatments; or the patient has received RAI treatments with a cumulative RAI dose of ≥22.2 GBq (600 mCi)

   Not a candidate for surgery or RAI therapy with curative intent.

   Lesions that would be treated by external beam radiation therapy (EBRT) based on standard of care can be so treated, but then cannot be used as target lesions.
2. Measurable disease by RECIST 1.1 criteria.
3. Documented disease progression by RECIST 1.1 in the past 14 months.
4. Availability of histological material (primary tumor or metastases) for review of the diagnosis and demonstration of PAX8-PPARgamma fusion gene.
5. Adequate TSH suppression (<0.5 mIU/L)
6. Prior chemotherapy or surgery must have been completed at least 28 days prior to registration, and all toxicities must have resolved.
7. Prior radioactive iodine must have been completed at least 6 months prior to registration, or there must be documented disease progression since such therapy if it was within 6 months. Sites that have received EBRT must have disease progression post-EBRT to be used as sites of measurable disease.
8. Life expectancy of greater than 6 months.
9. ECOG performance status 2 or less.
10. Patients must have normal organ function as defined below:

    AST(SGOT)/ALT(SGPT) less than 2.5 X institutional upper limit of normal (within 1 month of study Day 1)
11. Patients must be able to consume oral medications.
12. Women of childbearing potential must have a negative pregnancy test at baseline prior to receiving any study drug and must practice effective contraception while on study. (Pregnant or lactating patients are excluded).
13. All patients must sign an informed consent prior to enrollment.

Exclusion Criteria:

1. Patients may not be receiving any other investigational agents.
2. Patients with known untreated brain metastases.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to pioglitazone.
4. Diagnosis of diabetes mellitus or current therapy with any drugs used to treat diabetes mellitus, including but not limited to insulin, sulfonylureas, metformin, rosiglitazone (Avandia), and pioglitazone (Actos) within 14 days of study Day 1
5. Therapy with rosiglitazone (Avandia) or pioglitazone (Actos) at any time since the diagnosis of thyroid cancer.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congestive heart failure, unstable angina pectoris, or cardiac arrhythmias.
7. Pregnant women are excluded from this study because pioglitazone is a U.S. Food and Drug Administration Pregnancy Category C drug. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pioglitazone, breastfeeding should be discontinued if the mother is treated with pioglitazone.
8. No concurrent radiotherapy or chemotherapy may be given to the patient during the administration of the study drug.
9. Patients with uncontrolled malabsorption syndromes.
10. Patients with a history of congestive heart failure of any New York Heart Association class.
11. Any medical or psychiatric illness which, in the opinion of the principal investigator, would compromise the patient's ability to tolerate this treatment regimen.
12. Use of rifampin (strong CYP2C8 inducer) within 14 days of study Day 1.
13. Other current malignancy than the disease under study.
14. Grade 2 or worse edema within 14 days of study Day 1, per CTCAE v4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Koenig, MD, PhD, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - University of Colorado, Aurora, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Giordano TJ, Haugen BR, Sherman SI, Shah MH, Caoili EM, Koenig RJ. Pioglitazone Therapy of PAX8-PPARgamma Fusion Protein Thyroid Carcinoma. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1277-1281. doi: 10.1210/jc.2017-02533. PMID 29373711

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone Treatment: If eligible, subjects can participate in 1 or both parts of this study as follows:
  Part 1: In the initial main portion of the study subjects will receive 24 -28 weeks of therapy with pioglitazone at the dosage approved for the control of diabetes. Response will be evaluated per RECIST. Safety measure are outlined in the protocol including weekly weigh ins, calls, labs, exams, etc.
  Part 2: A secondary protocol is then available to subjects who complete the main initial study with less than complete response per RECIST. They can undergo a radioiodine scan to see if the treatment with pioglitazone has sensitized their disease to radioiodine. If it has - they can pursue the radioiodine treatment.
  Pioglitazone
Period: Overall Study
Arm/Group | Pioglitazone Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pioglitazone Treatment: Part 1: In the initial main portion of the study subjects will receive 24 -28 weeks of therapy with pioglitazone at the dosage approved for the control of diabetes. Response will be evaluated per RECIST. Safety measure are outlined in the protocol including weekly weigh ins, calls, labs, exams, etc.
Arm/Group | Pioglitazone Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response (Change)
Description: Response is measured by change in Tumor size (cm)
Time Frame: Baseline and 24 weeks
Measure: Number; unit: cm
Arm/Group | Pioglitazone Treatment
Number analyzed (Participants) | 1
cm
  Baseline | 6.0
  24 weeks | 3.9

2. Secondary Outcome: Change in Serum Thyroglobulin
Description: Determine if pioglitazone decreases serum thyroglobulin in patients with follicular-patterned thyroid carcinomas that contain the PAX8-PPARgamma fusion gene.
Time Frame: Baseline and 24 weeks
Measure: Number; unit: ng/mL
Arm/Group | Pioglitazone Treatment
Number analyzed (Participants) | 1
ng/mL
  Baseline | 1974
  24 weeks | 49.4

3. Secondary Outcome: Toxicity
Description: Toxicities experienced by patients with PAX8-PPARgamma fusion gene-positive follicular-patterned thyroid carcinomas treated with pioglitazone are indicated by presence of Serious Adverse Events (that show relatedness).
Time Frame: 24 weeks
Measure: Number; unit: serious adverse events
Arm/Group | Pioglitazone Treatment
Number analyzed (Participants) | 1
serious adverse events | 0

4. Other Pre Specified Outcome: Biomarkers
Description: Define predictive markers of response or insensitivity to pioglitazone. Unstained tumor tissue slides from archival paraffin blocks, fresh biopsy specimens from measurable metastases, and blood samples (serum and peripheral blood cells) will be collected on enrolled patients who consented for the optional correlative studies. These will be used to identify factors that predict efficacy of pioglitazone. Analyses may include measures of expression of specific RNAs and proteins, and DNA sequence analysis.
Time Frame: 24 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Sensitization to Radioiodine Therapy
Description: Determine if pioglitazone induces a clinically significant level of radioiodine uptake in the residual thyroid carcinoma, and if so, whether there is a therapeutic response to radioiodine. This will be addressed in a separate follow-up protocol available to subjects completing this study.
Time Frame: 24 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Lipid Accumulation in Tumor
Description: Determine (by MRI) if pioglitazone induces lipid accumulation in follicular-patterned thyroid carcinomas that contain the PAX8-PPARgamma fusion gene.
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Pioglitazone Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT01655719/Prot_SAP_000.pdf